CLINICAL TRIAL: NCT01416662
Title: Pharmacogenetics of Gemcitabine: Study of the Impact of Genetic Polymorphism of Cytidine Deaminase (CDA) on Toxicity in Resected Pancreatic Adenocarcinomas
Brief Title: Gemcitabine Hydrochloride in Treating Patients With Pancreatic Cancer That Has Been Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000703689; FFCD-1004; EU-21118; EUDRACT-2010-022987-11
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IA pancreatic cancer; stage IB pancreatic cancer; stage IIA pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine (Other): gemcitabine
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This clinical trial is studying gemcitabine hydrochloride in treating patients with pancreatic cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the ability of cytidine deaminase (CDA) to predict the occurrence of early (during the first 2 courses) severe hematological toxicity (grade 3 or 4), induced by gemcitabine hydrochloride in patients with resected pancreatic adenocarcinoma.

Secondary

* To determine the ability of CDA to predict the occurrence of severe non-hematological toxicity (grade 3 or 4), early (during the first 2 courses), and during the following courses, induced by gemcitabine hydrochloride.
* To determine the ability of CDA to predict the occurrence of severe hematological toxicity (grade 3 or 4) during all courses, induced by gemcitabine hydrochloride.
* To determine the impact of CDA status on gemcitabine hydrochloride pharmacokinetics and the ratio of gemcitabine hydrochloride/dFdU metabolization.
* To study genotype to phenotype of the CDA gene.
* To identify new mutations on the CDA gene.
* To evaluate the relationship between CDA status and global survival. (Exploratory)

OUTLINE: This is a multicenter study.

Within 8 weeks of resection, patients receive adjuvant gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacogenetic and biomarker studies. Some patients may undergo blood sample collection for pharmacokinetic studies.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * No metastatic or locally advanced (nonresectable) disease
* Must have undergone curative surgical resection

  * Must have macroscopically complete (R0 or R1) surgical outcome
* Adjuvant treatment with gemcitabine hydrochloride (for 6 months) is necessary, and able to start treatment within 8 weeks of surgical resection
* No ampullomas or endocrine carcinomas

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Alkaline phosphatases ≤ 5 times upper limit of normal
* Total bilirubin ≤ 50 µmol/L
* Creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Able to start adjuvant chemotherapy within 8 weeks of surgery
* No evolving infectious syndrome (fever > 38°C or abscess)
* No contraindication for gemcitabine hydrochloride
* No prior malignant tumor except for cutaneous basocellular carcinoma or in situ cervical epithelioma (prior history of malignant tumor diagnosed and treated more than 10 years ago allowed, except for breast cancer and melanoma)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No chemotherapy or radiotherapy within the past 10 years
* No prior ablation surgery leaving macroscopic tumor residues (R2)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
capability of CDA to predict the occurrence of early severe hematological toxicity upon gemcitabine | 2 months

SECONDARY OUTCOMES:
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Dahan, MD, Principal Investigator — CHU de la Timone
Locations (1):
- CHU de la Timone, Marseille, France

REFERENCES:
- [Result] Serdjebi C, Gagniere J, Desrame J, Fein F, Guimbaud R, Francois E, Andre T, Seitz JF, Monterymard C, Arsene D, Volet J, Abakar-Mahamat A, Lecomte T, Guerin-Meyer V, Legoux JL, Deplanque G, Guillet P, Ciccolini J, Lepage C, Dahan L. FFCD-1004 Clinical Trial: Impact of Cytidine Deaminase Activity on Clinical Outcome in Gemcitabine-Monotherapy Treated Patients. PLoS One. 2015 Aug 26;10(8):e0135907. doi: 10.1371/journal.pone.0135907. eCollection 2015. PMID 26308942